CLINICAL TRIAL: NCT00318357
Title: CARE-HF LTFU: CArdiac REsynchronization in Heart Failure Long-term Follow-up
Brief Title: CARE-HF Long Term Follow-up
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: CARE-HF Long-term follow-up
Record Dates: First submitted 2006-04-25; First posted 2006-04-26 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure
Keywords: Cardiac Resynchronization therapy (CRT); All-cause mortality; Long-term follow-up
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — No biospecimens are retained
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CRT in CARE-HF: In the CARE-HF study patients treated with standard medical treatment plus CRT were compared to patients treated with standard medical treatment. In the CARE-HF Long Term Follow-up part, all patients received CRT therapy on top of Optimal Medical Treatment. The CARE-HF LTFU study aims to further investigate mortality.
  CARE-HF LTFU study continued ot follow up the original CARE-HF CRT group patients.
  Interventions: Device: Continuation of CRT
- Control in CARE-HF: In the CARE-HF study patients treated with standard medical treatment. In the CARE-HF Long Term Follow-up part, almost all patients received CRT therapy on top of Optimal Medical Treatment. The CARE-HF LTFU study aims to further investigate mortality.
  CARE-HF LTFU study continued to follow up the original CARE-HF control group patients.
  Interventions: Device: Upgrade to CRT

INTERVENTIONS:
Device: Continuation of CRT — Implantation of CRT device and medical treatment according normal hospital routine.
  Other Names: Resynchronisation system of the InSync® family
  Groups: CRT in CARE-HF
Device: Upgrade to CRT — Recommended implantation of a Medtronic CRT InSync® family devices. Implantation of CRT device and medical treatment according normal hospital routine.
  Other Names: Resynchronisation system of the InSync® family
  Groups: Control in CARE-HF

SUMMARY:
The CARE-HF long-term follow-up trial evaluates the effects of cardiac resynchronization (CR) therapy on the mortality of patients from the CARE-HF program for an additional 4 year follow-up. Investigators are free to choose whatever available treatment they believe is in the patient's best interest.

DETAILED DESCRIPTION:
The CARE-HF study enrolled 813 patients from 82 centers in 12 European countries (Austria, Belgium, Denmark, Finland, France, Germany, Italy, Netherlands, Spain, Sweden, Switzerland, and UK). All patients that were reported to be alive in May 2005 will be asked to participate.

In the CARE-HF LTFU program patients from the CARE-HF trial were asked to be enrolled for an additional 4 year follow-up. Investigators were free to choose whatever available treatment they believe is in the patient's best interest, however the outcome of the CARE-HF trial suggested that all patients should receive CRT therapy on top of Optimal Medical Treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have participated in the CARE-HF program and were reported to be alive in May 2005
* Patients who signed a patient data release consent form

Exclusion Criteria:

* Patients who have not participated in the CARE-HF program
* Patients with exclusion criteria required by local legislation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic heart failure patients with NYHA class III-IV,with a LVEF of less than or equal to 35%, who are on optimal medical treatment, and documented evidence of ventricular dyssynchrony as evidenced by QRS or Echo prior enrollment in the CARE-HF main study.
  Patients who have participated in the CARE-HF program and were reported to be alive in May 2005 (study closure of the main study) are asked to participate in the CARE-HF LTFU study.
Sampling Method: Non-Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2006-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Cleland, Professor, Study Chair — The University of Hull; Department of Cardiology; United Kingdom
Locations (1):
- Hull Royal Infirmary - Academic Cardiology Unit, Cottingham, Kingston-Upon-Hull, United Kingdom

REFERENCES:
- [Background] Cleland JG, Daubert JC, Erdmann E, Freemantle N, Gras D, Kappenberger L, Klein W, Tavazzi L; CARE-HF study Steering Committee and Investigators. The CARE-HF study (CArdiac REsynchronisation in Heart Failure study): rationale, design and end-points. Eur J Heart Fail. 2001 Aug;3(4):481-9. doi: 10.1016/s1388-9842(01)00176-3. PMID 11511435
- [Result] Cleland JG, Daubert JC, Erdmann E, Freemantle N, Gras D, Kappenberger L, Tavazzi L; Cardiac Resynchronization-Heart Failure (CARE-HF) Study Investigators. The effect of cardiac resynchronization on morbidity and mortality in heart failure. N Engl J Med. 2005 Apr 14;352(15):1539-49. doi: 10.1056/NEJMoa050496. Epub 2005 Mar 7. PMID 15753115
- [Result] Cleland JG, Freemantle N, Erdmann E, Gras D, Kappenberger L, Tavazzi L, Daubert JC. Long-term mortality with cardiac resynchronization therapy in the Cardiac Resynchronization-Heart Failure (CARE-HF) trial. Eur J Heart Fail. 2012 Jun;14(6):628-34. doi: 10.1093/eurjhf/hfs055. Epub 2012 May 2. PMID 22552183

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient alive from original CARE-HF study consented for long term follow-up
Groups:
- Cardiac Resynchromization Therapy: In the CARE-HF study patients treated with standard medical treatment plus CRT were compared to patients treated with standard medical treatment.
  Medtronic CRT InSync® family devices : Implantation of CRT device and medical treatment according normal hospital routine.
- Cardiac Resynchromization Therapy (Control Pts in CARE-HF: In the CARE-HF study patients treated with standard medical treatment plus CRT were compared to patients treated with standard medical treatment. After release
  Medtronic CRT InSync® family devices : Implantation of CRT device and medical treatment according normal hospital routine.
Period: Overall Study
Arm/Group | Cardiac Resynchromization Therapy | Cardiac Resynchromization Therapy (Control Pts in CARE-HF
Started | 173 | 136
Completed | 134 | 104
Not Completed | 39 | 32

BASELINE CHARACTERISTICS:
Groups:
- Cardiac Resynchromization Therapy (Control Pts in CARE-HF): In the CARE-HF study patients treated with standard medical treatment. In the CARE-HF Long Term Follow-up part, almost all patients received CRT therapy on top of Optimal Medical Treatment. The CARE-HF LTFU study aims to further investigate mortality.
  CARE-HF LTFU study continued to follow up the original CARE-HF control group patients. With a recommended implantation of a Medtronic CRT InSync® family devices. Implantation of CRT device and medical treatment according normal hospital routine.
- Total: Total of all reporting groups
Arm/Group | Cardiac Resynchromization Therapy (Control Pts in CARE-HF) | Cardiac Resynchromization Therapy | Total
Number analyzed (Participants) | 136 | 173 | 309
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [56 to 70] | 65 [59 to 71] | 65 [56 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 45 | 84
  Male | 97 | 128 | 225
NYHA functional class III [Number; unit: participants] — New York Heart Association (NYHA) functional classification. It places patients in one of four catagories based on how much they are limited during physical activity. NYHA class III patient symptoms: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  participants | 132 | 165 | 297
QRS [Median (Inter-Quartile Range); unit: ms] | 160 [152 to 180] | 160 [152 to 180] | 160 [152 to 180]

OUTCOME MEASURES:

1. Primary Outcome: All Cause Mortality
Description: Long-term mortality with cardiac resynchronization therapy in the Cardiac Resynchronization-Heart Failure (CARE-HF) trial.
  The patients that were still alive after closure of the CARE-HF study (2005,NCT00170300), that were willing to participate in the CARE-HF LTFU study continued additional follow-up for 4 years, till end 2009. The reported mortality data is the combined mortality of the CARE-HF and the CARE-HF LTFU study. Study start CARE-HF 2000.
Time Frame: 8-year
Population: Data from the CARE-HF and CARE-HF Long-Term Follow-Up studies were combined for analysis
Measure: Number; unit: percentage of participants
Groups:
- Cardiac Resynchronization Therapy: In the CARE-HF study patients treated with standard medical treatment plus CRT were compared to patients treated with standard medical treatment.
  Medtronic CRT InSync® family devices : Implantation of CRT device and medical treatment according normal hospital routine.
- Upgrade to Cardiac Resynchronization Therapy: In the CARE-HF study patients treated with standard medical treatment. In the CARE-HF Long Term Follow-up part, almost all patients received CRT therapy on top of Optimal Medical Treatment. The CARE-HF LTFU study aims to further investigate mortality.
  CARE-HF LTFU study continued to follow up the original CARE-HF control group patients. With a recommended implantation of a Medtronic CRT InSync® family devices. Implantation of CRT device and medical treatment according normal hospital routine.
Arm/Group | Cardiac Resynchronization Therapy | Upgrade to Cardiac Resynchronization Therapy
Number analyzed (Participants) | 173 | 136
percentage of participants | 54.8 | 64.8
Statistical Analysis 1: Comparison: Cardiac Resynchronization Therapy vs Upgrade to Cardiac Resynchronization Therapy; Mortality is compared between the arms of the CARE-HF study, using Cox proportional hazards regression. Data from the original CARE-HF trial and the CARE-HF Long Term Follow-up trial were combined for the analysis; Test type: Superiority; p = 0.007, Regression, Cox

ADVERSE EVENTS:
Time Frame: 8-year. The patients that were still alive after closure of the CARE-HF study (2005,NCT00170300), that were willing to participate in the CARE-HF LTFU study continued additional follow-up for 4 years, till end 2009. The reported mortality data is the combined mortality of the CARE-HF and the CARE-HF LTFU study. Study start CARE-HF 2000.During the CARE-HFF LTFU study only mortality data was collected, no other adverse event data was collected..
Description: No Serious Adverse Events or Adverse events were collected during the CARE-HF LTFU study.
  All-Cause Mortality was monitored/assessed. Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Groups:
- Upgrade to Cardiac Resynchronization Therapy: CARE-HF LTFU study continued to follow up the original CARE-HF control group patients. With a recommended implantation of a Medtronic CRT InSync® family devices. Implantation of CRT device and medical treatment according normal hospital routine.
Arm/Group | Cardiac REsynchronization Therapy | Upgrade to Cardiac Resynchronization Therapy
All-Cause Mortality (participants affected / at risk) | 39/173 | 32/136
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days